CLINICAL TRIAL: NCT00126607
Title: Phase II Study of Trastuzumab (NSC-688097) in Advanced High Grade Salivary Gland Carcinoma
Brief Title: Trastuzumab in Treating Patients With Metastatic or Recurrent Salivary Gland Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03172; S0431; U10CA032102 (NIH); CDR0000437831 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: High-grade Salivary Gland Mucoepidermoid Carcinoma; Recurrent Salivary Gland Cancer; Salivary Gland Acinic Cell Tumor; Salivary Gland Adenocarcinoma; Salivary Gland Poorly Differentiated Carcinoma; Stage IVA Salivary Gland Cancer; Stage IVB Salivary Gland Cancer; Stage IVC Salivary Gland Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Trastuzumab

ARMS (1):
- Treatment (trastuzumab) (Experimental): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well trastuzumab works in treating patients with metastatic or recurrent salivary gland cancer. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess response (confirmed and unconfirmed, complete and partial response) in patients with advanced high-grade salivary gland carcinoma treated with trastuzumab.

II. To assess one-year progression-free survival and one-year overall survival for patients treated with this regimen.

III. To assess the toxicities associated with this treatment regimen in this group of patients.

IV. To measure the indicators of C-erb B2 oncoprotein expression and C-erb B2 oncogene amplification and epidermal growth factor receptor expression and explore the relationship between these markers and response, progression-free survival and overall survival in preliminary fashion.

OUTLINE: Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 8 weeks until disease progression and then every 3 months for 1 year and every 6 months until 3 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant high-grade (poorly differentiated or undifferentiated) salivary gland carcinoma of the head and neck (except adenoid cystic carcinoma) that is either metastatic or recurrent and is not amenable to salvage surgical resection or radiation therapy; eligible histologies are adenocarcinoma, acinic cell carcinoma, mucoepidermoid carcinoma, salivary duct carcinoma and undifferentiated carcinoma
* Patients must have tumors that car HER-2 gene amplification as determined by (i) fluorescence in situ hybridization (FISH) or (ii) overexpression of HER-2 protein, 2+ to 3+ level assessed by immunohistochemistry
* Patients must have measurable disease; all measurable disease must be assessed within 28 days prior to registration; all non-measurable disease must be assessed within 42 days prior to registration
* Patients with known brain metastases are not eligible for this trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients must have and must be willing to submit tumor tissue for pathology review and translational medicine studies; patients must be offered the opportunity to participate in specimen banking for future research
* Patients previously treated with chemotherapy are eligible provided that at least (28 days) has elapsed since the last course of chemotherapy was completed and patient has recovered from all toxicities
* Prior radiation must have been completed at least 28 days prior to registration and all toxicities must have resolved (in the opinion of the treating investigator); prior surgery must have been completed at least 28 days prior to registration and all surgical adverse events must have resolved (in the opinion of the treating investigator)
* Patients must not be planning on receiving any other investigational agents, other chemotherapeutic agents, radiation therapy, or hormonal therapy while receiving treatment on this study except for steroids administered for non-disease-related conditions (e.g., insulin for diabetes)
* Patients must have a Zubrod Performance status of 0-2
* WBC count >= 2,000 ul within 28 days prior to registration
* ANC count >= 1,000/ul within 28 days prior to registration
* Platelet count >= 75,000/ul within 28 days prior to registration
* Bilirubin =< 2.5 x the institutional upper limit of normal within 28 days prior to registration
* SGOT or SGPT =< 2.5 x the institutional upper limit of normal within 28 days prior to registration
* Patients with liver metastases must have bilirubin and SGOT or SGPT =< 5 x the institutional upper limit of normal
* Serum creatinine < 2.5 x the institutional limit of normal within 28 days prior to registration
* Patients with a known history of allergic reactions to compounds of similar chemical or biologic composition to trastuzumab are not eligible
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day
* In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the data operations center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-07; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response (confirmed and unconfirmed, complete and partial response) in patients treated with trastuzumab | Up to 4 years
  A true response probability of 30% or greater would be of interest.

SECONDARY OUTCOMES:
Progression-free survival | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 1 year
Overall survival | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Kane, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States